CLINICAL TRIAL: NCT06207747
Title: Quantitative Analysis of PET/CT Images of Immune Related Side Effects in Metastatic Melanoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KME RS 0120-256/2020-14
Record Dates: First submitted 2023-12-28; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-11

CONDITIONS: Melanoma; PET CT
Keywords: PET/CT; melanoma; immunotherapy; side-effects
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: This study will prospectively collect data from metastatic or stage III.D unresectable melanoma patients treated with ICIs and followed regularly with 18F-FDG PET/CT scans. Recruitment is expected to last 18 months. Predictive sample size is 100 melanoma patients.
  Timing of PET/CT scans:
  * Baseline PET/CT less than 4 weeks before first ICI infusion
  * Follow-up: 4 weeks (+/- 5 days) after first infusion, 16 weeks (+/- 7 days) after first infusion, then after every 16 weeks (+/- 7 days) or before in case of PD suspicion .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This study will prospectively collect data from metastatic or stage III.D unresectable melanoma pts (Experimental): Timing of PET/CT scans:
  * Baseline PET/CT less than 4 weeks before first ICI infusion
  * Follow-up: 4 weeks (+/- 5 days) after first infusion, 16 weeks (+/- 7 days) after first infusion, then after every 16 weeks (+/- 7 days) or before in case of PD suspicion
  Interventions: Diagnostic Test: additional PET/CT at 4 weeks, analysing using quantative analysis

INTERVENTIONS:
Diagnostic Test: additional PET/CT at 4 weeks, analysing using quantative analysis — Patient with metastatic melanoma will be monitored with additional PET/CT at 4 weeks, analysing using quantative analysis will be done.

SUMMARY:
New cancer treatment with immune-checkpoint inhibitors (ICIs) has changed the way patients with melanoma and a variety of other cancers are being treated. Many pivotal trials that showed efficacy and safety of ICIs were performed in malignant melanoma. ICI can cause a different type of toxicity, called immune-related adverse events (irAEs). Though the exact pathophysiology is not completely understood, it is believed that irAEs are provoked by immune upregulation and inflammation. However, they can be serious, life-threatening, and warrant hospital admission as well. Dangerous irAEs include myocarditis, myositis, and pneumonitis, among others. Due to the novel mechanism of action, unpredictable nature, and wide usage of this type of treatment in the future, there is urgent need for better control of these potentially dangerous side effects. Early recognition and treatment of irAEs are of great importance in successful management.

Positron emission tomography-computed tomography (PET/CT) with [18F]2fluoro-2-deoxy-D-glucose (18F-FDG) is a sensitive, non-invasive, and widely used method for diagnosis and evaluation of treatment efficacy of malignant melanoma. The combination of 18F-FDG-PET and CT allows for assessment of both functional and morphological status of the lesions, and so facilitates better clinical decisions and patient care during treatment. It is also a very sensitive method for recognising inflammation, that can be a signal of irAEs.

Quantitative analysis is a rapidly evolving field of PET/CT image analysis. It includes both radiomics and artificial intelligence. Some studies have reported that quantitative analysis could predict efficacy of different cancer treatments. Quantitative image analysis in cancer response assessment is a rapidly expanding field, with the ultimate goal of clinical translation. However, in the specific instance of irAE diagnosis, it is not yet clear what role quantitative analysis of PET/CT scans can play.

The hypothesis is that quantitative analysis of PET/CT images provides more information on possible irAE, thus helping to treat these side effects more quickly and successfully.

DETAILED DESCRIPTION:
New cancer treatment with immune-checkpoint inhibitors (ICIs) has changed the way patients with melanoma and a variety of other cancers are being treated. Based on many positive randomised controlled trials in metastatic and neo-/adjuvant setting, ICI agents targeting programmed death-1 (PD-1), programmed death ligand-1 (PD-L1) and cytotoxic T-lymphocyte antigen-4 (CTLA-4) have become invaluable in the treatment of different carcinomas. Many pivotal trials that showed efficacy and safety of ICIs were performed in malignant melanoma.

ICI can cause a different type of toxicity, called immune-related adverse events (irAEs), that can occur in any organ of the body. Though the exact pathophysiology is not completely understood, it is believed that irAEs are provoked by immune upregulation and inflammation. In general, they are less frequent compared to chemotherapy toxicities and usually low grade and manageable. However, they can be serious, life-threatening, and warrant hospital admission as well. Dangerous irAEs include myocarditis, myositis, and pneumonitis, among others. Due to the novel mechanism of action, unpredictable nature, and wide usage of this type of treatment in the future, there is urgent need for better control of these potentially dangerous side effects. Early recognition and treatment of irAEs are of great importance in successful management.

Positron emission tomography-computed tomography (PET/CT) with [18F]2fluoro-2-deoxy-D-glucose (18F-FDG) is a sensitive, non-invasive, and widely used method for diagnosis and evaluation of treatment efficacy of malignant melanoma. The combination of 18F-FDG-PET and CT allows for assessment of both functional and morphological status of the lesions, and so facilitates better clinical decisions and patient care during treatment. It is also a very sensitive method for recognising inflammation, that can be a signal of irAEs.

Quantitative analysis is a rapidly evolving field of PET/CT image analysis. It includes both radiomics and artificial intelligence. Quantitative analyses of medical images provide insight into hidden information about the image, which is usually not fully assessed by a nuclear medicine specialist (for example, information on the spatial heterogeneity of the tumour). Some studies have reported that quantitative analysis could predict efficacy of different cancer treatments. Quantitative image analysis in cancer response assessment is a rapidly expanding field, with the ultimate goal of clinical translation. However, in the specific instance of irAE diagnosis, it is not yet clear what role quantitative analysis of PET/CT scans can play.

The hypothesis is that quantitative analysis of PET/CT images provides more information on possible irAE, thus helping to treat these side effects more quickly and successfully. The association of quantitative PET/CT analysis with patient survival and the predictive value of an early-time point PET/CT scan in response to ICIs will be prospectively examined. The positive impact or irAE of autoimmune thyroiditis on the outcome of ICIs treatment will be also will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* - Older than 18 years old
* Cyto- or histologically proven melanoma
* Stage III.D unresectable/ stage IV melanoma (AJCC classification, 8th edition, 2018)
* Asymptomatic brain metastases
* Three measurable metastatic lesions
* 1st, 2nd, further line of systemic treatment with ICIs (either ipilimumab, nivolumab, pembrolizumab, or combination)
* PS WHO 0-2 (ECOG criteria)
* FDG-PET within four weeks of treatment initiation
* Written consent form

Exclusion Criteria:

* Symptomatic brain metastases
* PS WHO > 2 (ECOG criteria)
* Contraindications for ICI treatment
* Other malignant diseases (not included: BCC, SCC, in situ carcinoma of cervix, other cured malignant diseases without relapse more than three years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
predictive value of PET/CT for detecting irAE | two years
  PET/CT will be performed regularly in metastatic melanoma patients treated with ICIs. Imaging will be analysed for detection of irAE, using in-depth radiological (nuclear) and quantitative (radiomic and artificial intelligence) analysis of affected organs. SUV percentiles of 18F-FDG uptake in the affected organs will be used for prediction of irAE.

CONTACTS AND LOCATIONS:
Overall Officials: Nežka Hribernik, M.D., Principal Investigator — Institute of Oncology Ljubljana, Slovenia
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hribernik N, Huff DT, Studen A, Zevnik K, Klanecek Z, Emamekhoo H, Skalic K, Jeraj R, Rebersek M. Quantitative imaging biomarkers of immune-related adverse events in immune-checkpoint blockade-treated metastatic melanoma patients: a pilot study. Eur J Nucl Med Mol Imaging. 2022 May;49(6):1857-1869. doi: 10.1007/s00259-021-05650-3. Epub 2021 Dec 27. PMID 34958422
- [Result] Huff DT, Ferjancic P, Namias M, Emamekhoo H, Perlman SB, Jeraj R. Image intensity histograms as imaging biomarkers: application to immune-related colitis. Biomed Phys Eng Express. 2021 Sep 30;7(6):10.1088/2057-1976/ac27c3. doi: 10.1088/2057-1976/ac27c3. PMID 34534974